CLINICAL TRIAL: NCT06048939
Title: Combined Effect of Aerobic and Resistance Training on Physical, Menstrual and Psychological Health of Adolescent Girls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01543 Saira Shabbir
Record Dates: First submitted 2023-07-23; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Psychological Well-Being
Keywords: psychological well-being; Menstrual Problem; Physical inactivity
MeSH Terms: conditions — Psychological Well-Being; Menstruation Disturbances; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic and resistance training (Experimental): moderate intensity aerobic and body weight resistance training on female adolescents.
  Interventions: Other: moderate intensity aerobic training and body weight resistance training
- aerobic training (Active Comparator): moderate intensity aerobic and body weight resistance training on female adolescents.
  Interventions: Other: moderate intensity aerobic training

INTERVENTIONS:
Other: moderate intensity aerobic training and body weight resistance training — Bodyweight Resistance exercises Frequency: twice a week Intensity: moderate Time: 40 Minutes Warm up: 10mins Rotations and Dynamic stretches Body weight resistance Exercises: 20mins Calf raises (1 x 10-15 Reps) Squats (1 x 10-15 Reps) Lunges (1 x 10-15 Reps on each side) Modified push-ups (1 x 10-15 Reps) Bridging (1 x 10-15 Reps) Plank hold (10 Seconds) Side planks (10 Seconds each side) Cool down: 10 mins Slow marching and static stretches for next 6 weeks progression will be made by adding one more set of same exercises Aerobic training: Frequency: 2 Days per week Intensity: 60% of maximum heart rate. Time: 45 Minutes Exercise Protocol Warm up: 10mins Rotations and Dynamic stretches
  Aerobic exercises will be same as given to control group
  Arms: aerobic and resistance training
Other: moderate intensity aerobic training — Aerobic Exercises Frequency: 2 Days per week Intensity: 60% of maximum heart rate. Time: 45 Minutes Warm up: 10mins Rotations and Dynamic stretches Aerobic exercises: 25 mins
  (1 minute of each exercise with 60 seconds rest and repeating the same sequence for 1 minute.) Exercises will be performed at slow pace Marching, Single step touch, Step touches front and back, Double step touch, "V" step, knee lift, leg curl , forward walk, reach outs, lunge side and back, "L" Step, jumping jacks Cool down: 10 mins Slow marching and static stretches for next 6weeks progression will be made by increasing speed of same exercises
  Arms: aerobic training

SUMMARY:
This study proposes to find out the Combined Effect of Aerobic & Resistance Training on physical, menstrual and psychological health of Adolescent Girls. The study results will be helpful to explore the mode and intensity of aerobic and resistance exercise and for creating strategies for improving the lifestyle of the adolescents by adopting the appropriate exercise guidelines.

DETAILED DESCRIPTION:
Adolescence is a time of rapid growth and development as well as a crucial time for the formation of behaviors connected to one's health (1). This stage is characterized by simultaneous hormonal, psychological, and physical changes. Regular exercise is an essential part of an all-encompassing plan to protect against numerous risk factors Physical inactivity, sedentary behavior and low cardio respiratory fitness are strong risk factors for morbidity and mortality. There is emerging evidence to link increased time spent using screens for leisure, with poorer mental health experiences among adolescents. Research has shown that physical activity can play a vital role in improving both their physical and psychological well-being.

The evidence suggests that moderate aerobic exercise can have a positive impact on menstrual cycle regularity and reducing menstrual pain. Resistance training can increase the levels of various hormones and neurotransmitters like endorphins, dopamine, serotonin, and nor epinephrine in the brain that are attributed to improved mood and reduced feelings of anxiety.

Aerobic exercise is performed by repeating sequences of light-to-moderate intensity activities for extended periods of time. Exercises are typically done at 60-70% of heart rate, while resistance training, also known as strength training, uses external resistance to enhance muscle mass, strength, tone, balance, and mental well-being Previous studies show that engaging adolescents in resistance or combined training is essential to the maintenance and/or improving muscular fitness. Another study reported both HIIT and MICT appear to be similarly effective on risk factors of CVD. Incorporating diverse exercises in physical education classes for adolescent girls improves overall fitness, benefiting their long-term health and well-being. The 2017 study highlighted the importance of expert trainers, supervision, and customized weight training in resistance training for children and adolescents, leading to improved physical fitness. Regular physical activity can reduce leptin levels and relax abdominal muscles, leading to pain relief and enhanced quality of life. Ginger, aerobic exercise, and stretching exercises can alleviate physical symptoms and reduce pain intensity and duration in girls with dysmenorrhea by promoting blood flow and metabolism in the uterus. Regular aerobic exercise reduces negative mood states and physical symptoms in women during the menstrual cycle, consistent with previous studies.

Aerobic exercise alleviates dysmenorrhea symptoms by releasing natural painkillers and suppressing the release of pain-causing prostaglandins during menstruation. Aerobic exercise may help reduce menstrual pain by increasing blood flow to working muscles, potentially relieving congestion.

Evidence demonstrates that menstrual cycle irregularity, which is most frequently addressed in adolescence, is also linked to sedentary lifestyle, psychological stress, and aggressive physical activity. There is a tonne of data that aerobic and resistance training affects vascular function, obesity, and diabetes.

The lack of research on the effects of aerobic and resistance training on adolescent girls' physical fitness, mental health, and menstrual cycle underscores the importance of understanding how physical activity influences these variables. A study found that Resistance band training for 8 weeks improved mood, behavior, and physical menstrual symptoms in non-athletic teenage girls with premenstrual syndrome. A study found that participating in an 8-week aerobic exercise program significantly reduced dysmenorrhea severity in medical students compared to a control group, as observed in the first and second menstrual cycles after the intervention. A study conducted in 2022 by a medical student found that vigorous exercise during menstruation can lead to increased estrogen and progesterone levels, resulting in more menstrual pain due to increased blood flow.

Evidence shows irregularity in menstrual cycle addressed most commonly in adolescents is associated with sedentary life style and psychological stress. The idea that exercise might help to relieve menstrual pain is not new. Aerobic exercise is one of the exercise option whose significant effects were seen in dysmenorrhea and pre-menstural symptoms. Gap regarding relief in menstrual cycle symtopms with resistance exercises is need to be filled. Furthermore no such study was done to compare the effects of aerobic and resistance exercises on menstrual, physical and psychological health of adolescent girls at a time. Therefore current study proposes to find out the Combined Effect of Aerobic & Resistance Training on these problems of Adolescent Girls. The study results will be helpful to explore the mode and intensity of resistance exercise and for creating strategies for improving the lifestyle of the adolescents by adopting the appropriate exercise guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescents who have achieved Menarche.
* 13-19 years of age
* BMI criteria: 17.50 - 22.99 (BMI Asia)
* Score less than 13 on IPAQ (Inactive)

Exclusion Criteria:

* History of musculoskeletal trauma or injury
* Any diagnosed psychological condition
* Participated in Exercise program for past 6 months

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Menstrual Health Instrument (MHI) | at 1st week and after 12th week
  The Menstrual Health Instrument (MHI) is a comprehensive 29-item scale that assesses the physical and emotional well-being of adolescents regarding menstruation. It covers five sub-scales and utilizes a 5-point Likert scale (from strongly disagree to strongly agree)

SECONDARY OUTCOMES:
The Alpha Health Related Fitness Test Battery for Children And Adolescents | at 1st week and after 12th week
  The Alpha Health Related Fitness Test Battery has been shown to have good validity in assessing health-related fitness components in children and adolescents. The results consistently demonstrate significant correlations, indicating that the test battery accurately measures these fitness components.

CONTACTS AND LOCATIONS:
Overall Officials: summra andleeb, MS(OMPT), Principal Investigator — riphah internation university
Locations (1):
- Vega school system Dinga, Dinga, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No